CLINICAL TRIAL: NCT04234464
Title: A Randomized, Double-blind, Single-dose, 2-Period, Crossover Study to Assess the Efficacy of PT027 Compared With Placebo on Exercise-Induced Bronchoconstriction in Adult and Adolescent Subjects With Asthma
Brief Title: A Study to Assess the Efficacy of Budesonide/Albuterol Metered-dose Inhaler (BDA MDI/PT027) on Exercise-induced Bronchoconstriction in Adults and Adolescents With Asthma
Acronym: TYREE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bond Avillion 2 Development LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV005
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Results first posted 2021-12-30 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Exercise Induced Bronchospasm
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A/B - Treatment with BDA MDI 160/180 followed by treatment with Placebo MDI (Experimental): Subjects randomized to receive a single dose of BDA MDI 160/180 in treatment period 1, and a single dose of Placebo MDI in treatment period 2.
  Interventions: Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg; Combination Product: Placebo metered-dose inhaler
- B/A - Treatment with Placebo MDI followed by treatment with BDA MDI 160/180 (Experimental): Subjects randomized to receive a single dose of Placebo MDI in treatment period 1, and a single dose of BDA MDI 160/180 in treatment period 2.
  Interventions: Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg; Combination Product: Placebo metered-dose inhaler

INTERVENTIONS:
Combination Product: Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg — Budesonide/albuterol sulfate combination inhalation aerosol single dose
  Other Names: BDA MDI 160/180 μg (PT027)
Combination Product: Placebo metered-dose inhaler — Placebo inhalation aerosol single dose
  Other Names: Placebo MDI

SUMMARY:
This is a multicenter, randomized, double-blind, single-dose, placebo-controlled, 2-period, crossover study to evaluate the efficacy and safety of budesonide/albuterol metered-dose inhaler (BDA MDI/PT027) as compared with a placebo metered-dose inhaler (placebo MDI) on exercise-induced bronchoconstriction (EIB) in adult and adolescent subjects with asthma. Subjects will receive each study treatment on separate visits and undergo a treadmill exercise challenge test for up to 10 minutes so that the effect of study treatment on exercise-induced bronchoconstriction can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 12 to 70 years at the time of informed consent
2. Documented history of asthma for at least 6 months prior to Visit 1
3. Receiving 1 of the following asthma therapies with stable dosing for at least the 4 weeks before Visit 1; no other asthma therapies are permitted during the study:

   * Short/rapid-acting β 2-adrenoreceptor agonist (SABA) used as needed
   * Low- to medium-dose maintenance therapy with inhaled corticosteroid (ICS) and SABA used as needed
4. Demonstrate acceptable MDI administration technique (use of a spacer device during the treatment phase is not permitted)

Exclusion Criteria:

1. Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia), including regular or occasional use of oxygen
2. Systemic corticosteroids (SCS) use (any dose and any indication) within 3 months before Visit 1
3. History of life-threatening asthma, defined by past intubations for asthma, or intensive care unit admission for asthma within the prior 24 months
4. Receiving regular maintenance treatment with prohibited anti-inflammatory or long-acting bronchodilator asthma medication (inhaled, nebulized, oral, or systemic) within 1 month prior to Visit 1
5. Unable to tolerate the lung function testing performed after exercise challenge test without use of rescue medication
6. Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months before Visit 1 (including all forms of tobacco, e-cigarettes [vaping], and marijuana)
7. Completed treatment for lower respiratory infection within 6 weeks prior to Visit 1, regardless if resulting in accompanying asthma symptoms aggravation or not
8. Upper respiratory infection involving antibiotic treatment not resolved within 7 days prior to Visit 1
9. Received any marketed (eg, omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab) or investigational biologic within 3 months before Visit 1, or any other prohibited medication
10. Current treatment with any investigational product or within the last 30 days of Visit 1.
11. Historical or current evidence of a clinically significant disease
12. Cancer not in complete remission for at least 5 years before Visit 1
13. Hospitalization for psychiatric disorder or attempted suicide within 1 year of Visit 1
14. History of psychiatric disease or intellectual deficiency
15. Having a scheduled or planned hospitalization during the study
16. Inability (and/or unwillingness) to abstain from protocol-defined prohibited medications during the study.
17. Use of any herbal products by inhalation or nebulizer within 2 weeks of Visit 1 and/or the unwillingness to stop during the study duration.
18. Significant abuse of alcohol or drugs

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Albers, MD, PhD, Study Director — Avillion LLP
Locations (6):
- United States (6):
  - Research Site, Denver, Colorado
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Skillman, New Jersey
  - Research Site, Raleigh, North Carolina
  - Research Site, Burke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] LaForce C, Chipps BE, Albers FC, Reilly L, Johnsson E, Andrews H, Cappelletti C, Maes A, Papi A. Albuterol/budesonide for the treatment of exercise-induced bronchoconstriction in patients with asthma: The TYREE study. Ann Allergy Asthma Immunol. 2022 Feb;128(2):169-177. doi: 10.1016/j.anai.2021.10.020. Epub 2021 Oct 24. PMID 34699967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects included in the study were male and female adults and adolescents 12 to 70 years of age with a diagnosis of asthma as defined by the Global Initiative for Asthma (GINA) criteria and EIB as defined by a >=20% decrease from pre-exercise challenge best FEV₁ observed within 60 minutes after an exercise challenge at both screening visits. The first subject enrolled on 15 January 2020 and the last subject completed the study on 28 August 2020. Subjects were enrolled at 6 US study centers.
Pre-assignment Details: The randomized treatment phase started after a 1 to 2 week screening period (Visits 1 and 2). In addition to the 60 subjects randomized, 71 subjects were screened but did not participate (70 screen failures, 1 withdrawal by subject).
Groups:
- A/B - Treatment With BDA MDI 160/180 Followed by Treatment With Placebo MDI: Subjects randomized to receive a single dose of BDA MDI (PT027) at Visit 3/Period 1, and a single dose of placebo MDI at Visit 4/Period 2.
  Visit 3/Period 1 (Day 1) - Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg: Budesonide/albuterol sulfate combination inhalation aerosol single dose.
  Visit 4/Period 2 (Day 8 +/- 6 days) - Placebo metered-dose inhaler: Placebo inhalation aerosol single dose.
- B/A - Treatment With Placebo MDI Followed by Treatment With BDA MDI 160/180: Subjects randomized to receive a single dose of placebo MDI at Visit 3/Period 1, and a single dose of BDA MDI (PT027) at Visit 4/Period 2.
  Visit 3/Period 1 (Day 1) - Placebo metered-dose inhaler: Placebo inhalation aerosol single dose.
  Visit 4/Period 2 (Day 8 +/- 6 days) - Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg: Budesonide/albuterol sulfate combination inhalation aerosol single dose.
Period: Period 1 (First Treatment Intervention)
Arm/Group | A/B - Treatment With BDA MDI 160/180 Followed by Treatment With Placebo MDI | B/A - Treatment With Placebo MDI Followed by Treatment With BDA MDI 160/180
Started | 29 | 31
Completed | 29 | 31
Not Completed | 0 | 0
Period: Period 2 (Second Treatment Intervention)
Arm/Group | A/B - Treatment With BDA MDI 160/180 Followed by Treatment With Placebo MDI | B/A - Treatment With Placebo MDI Followed by Treatment With BDA MDI 160/180
Started | 29 | 31
Completed | 28 | 31
Not Completed | 1 | 0
Not completed — Subject did not meet the pre-dose FEV₁ criterion of >70% predicted at Visit 4/Visit 4 repeat. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- A/B - Treatment With BDA MDI 160/180 Followed by Treatment With Placebo MDI: Subjects randomized to receive single dose of BDA MDI (PT027) at Visit 3/Period 1, and a single dose of placebo MDI at Visit 4/Period 2.
  Visit 3/Period 1 (Day 1) - Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg: Budesonide/albuterol sulfate combination inhalation aerosol single dose
  Visit 4/Period 2 (Day 8 +/- 6 days) - Placebo metered-dose inhaler: Placebo inhalation aerosol single dose
- B/A - Treatment With Placebo MDI Followed by Treatment With BDA MDI 160/180: Subjects randomized to receive single dose of placebo MDI at Visit 3/Period 1, and a single dose of BDA MDI (PT027) at Visit 4/Period 2.
  Visit 3/Period 1 (Day 1) - Placebo metered-dose inhaler: Placebo inhalation aerosol single dose
  Visit 4/Period 2 (Day 8 +/- 6 days) - Budesonide/albuterol sulfate metered-dose inhaler 160/180 μg: Budesonide/albuterol sulfate combination inhalation aerosol single dose
- Total: Total of all reporting groups
Arm/Group | A/B - Treatment With BDA MDI 160/180 Followed by Treatment With Placebo MDI | B/A - Treatment With Placebo MDI Followed by Treatment With BDA MDI 160/180 | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 27 | 30 | 57
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.28) | 41.8 (11.31) | 40.5 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 29 | 28 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 13 | 18
  White | 21 | 18 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 60
Height [Mean (Standard Deviation); unit: Centimeters] | 167.0 (9.41) | 170.7 (10.28) | 168.9 (9.96)
Weight [Mean (Standard Deviation); unit: Kilograms] | 81.3 (18.50) | 84.4 (21.60) | 82.9 (20.05)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per meter squared] | 29.0 (5.51) | 28.7 (5.52) | 28.8 (5.47)
Maximal Heart Rate at Screening Visit 1 [Mean (Standard Deviation); unit: Beats per minute] | 167.2 (15.11) | 164.1 (12.71) | 165.6 (13.90)
Maximal Heart Rate at Screening Visit 2 [Mean (Standard Deviation); unit: Beats per minute] | 166.3 (15.83) | 163.3 (12.88) | 164.8 (14.34)
Pre-dose pre-ECT FEV₁ [Mean (Standard Deviation); unit: Liters] | 2.712 (0.5895) | 2.608 (0.6409) | 2.658 (0.6137)
Pre-dose pre-ECT FEV₁ % predicted normal [Mean (Standard Deviation); unit: Percentage of predicted normal] | 84.86 (12.914) | 78.24 (6.567) | 81.44 (10.593)
Pre-dose pre-ECT FVC [Mean (Standard Deviation); unit: Liters] | 3.823 (0.9770) | 3.546 (1.0576) | 3.680 (1.0204)
Pre-dose pre-ECT FEV₁/FVC [Mean (Standard Deviation); unit: Percent] | 71.88 (8.143) | 74.97 (9.051) | 73.47 (8.692)
Time since diagnosis of asthma to randomization [Median (Full Range); unit: years] | 25.19 [2.5 to 54.6] | 28.59 [3.4 to 56.1] | 27.36 [2.5 to 56.1]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percentage Fall From Post-dose, Pre-exercise Baseline in Forced Expiratory Volume in 1 Second (FEV₁) Observed up to 60 Minutes Post-exercise Challenge
Description: Lung function was measured by spirometry. Spirometry assessments were completed 5 minutes before dosing, 30 minutes after dosing (baseline; 5 minutes before the exercise challenge), and then 5, 10, 15, 30, and 60 minutes after the exercise challenge. A reduction in FEV₁ was expected due to the effects of asthma and exercise on breathing and lung function. The percentage fall in FEV₁ was calculated based on the baseline value and maximum percentage fall value during the 60-minute assessment period.
Time Frame: Up to 60 minutes post exercise challenge
Measure: Least Squares Mean (95% Confidence Interval); unit: Maximum percentage fall FEV₁
Groups:
- Treatment Intervention A - BDA MDI 160/180 - All Subjects: Analysis of subjects receiving Treatment Intervention A - BDA MDI 160/180
- Treatment Intervention B - Placebo MDI - All Subjects: Analysis of subjects receiving Treatment Intervention B - Placebo MDI
Arm/Group | Treatment Intervention A - BDA MDI 160/180 - All Subjects | Treatment Intervention B - Placebo MDI - All Subjects
Number analyzed (Participants) | 60 | 59
Maximum percentage fall FEV₁ | 5.45 [2.56 to 8.35] | 18.97 [16.06 to 21.88]
Statistical Analysis 1: Comparison: Treatment Intervention A - BDA MDI 160/180 - All Subjects vs Treatment Intervention B - Placebo MDI - All Subjects; Maximum percentage fall in post-dose pre-exercise FEV₁ up to 60 minutes post-exercise challenge is analyzed using a mixed effects model adjusted for treatment, treatment period, treatment sequence as categorical fixed effects, period-specific pre-dose baseline FEV₁ and average pre-dose baseline FEV₁ as continuous covariates, and a random subject within treatment sequence effect; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 13.51, 95% CI 2-sided [10.09 to 16.94]

2. Secondary Outcome: Percentage of Subjects With a Maximum Percentage Fall in FEV₁ Post-exercise Challenge of <10%
Description: The percentage fall in FEV₁ was calculated based on the baseline value and maximum percentage fall value during the 60-minute assessment period, and the percentage of subjects with a maximum percentage fall <10% was determined.
Time Frame: Up to 60 minutes post exercise challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Intervention A - BDA MDI 160/180 - All Subjects | Treatment Intervention B - Placebo MDI - All Subjects
Number analyzed (Participants) | 60 | 60
Participants | 47 | 17
Statistical Analysis 1: Comparison: Treatment Intervention A - BDA MDI 160/180 - All Subjects vs Treatment Intervention B - Placebo MDI - All Subjects; A generalized linear mixed model with logit link adjusted for treatment, treatment period and treatment sequence as fixed effects, pre-dose baseline FEV₁ and average pre-dose baseline FEV₁ as continuous covariates, and a random subject within treatment sequence effect; Test type: Superiority; p < 0.001, Mixed Models Analysis; Odds Ratio (OR) = 10.548, 95% CI 2-sided [4.311 to 25.805]

ADVERSE EVENTS:
Time Frame: Approximately one week for each treatment intervention.
Description: Safety population included all subjects who received at least one treatment intervention.
Groups:
- Treatment Intervention - BDA MDI 160/180 - All Subjects: Safety analysis of subjects receiving Treatment A - BDA MDI 160/180
- Treatment Intervention - Placebo MDI - All Subjects: Safety analysis of subjects receiving Treatment B - Placebo MDI
Arm/Group | Treatment Intervention - BDA MDI 160/180 - All Subjects | Treatment Intervention - Placebo MDI - All Subjects
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 2/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Intervention - BDA MDI 160/180 - All Subjects (N=60) | Treatment Intervention - Placebo MDI - All Subjects (N=59)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data or results obtained from this study must not be published without prior approval from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04234464/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT04234464/SAP_001.pdf